CLINICAL TRIAL: NCT05287243
Title: The Impact of a Customized Respiratory Muscle Training and Maintenance Program on Cardiopulmonary Function in People With Parkinson's Disease.
Brief Title: Impact of Customized Respiratory Training on Cardiopulmonary Function in Parkison's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of St. Augustine for Health Sciences (Other)
Responsible Party: Principal Investigator, Kristen Barta, Associate Professor, University of St. Augustine for Health Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PT-0928-306
Record Dates: First submitted 2022-03-10; First posted 2022-03-18 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inspiratory Muscle Training (Other): involves the intervention portion of the study to improve strength of the cardiopulmonary system
  Interventions: Other: inspiratory muscle training

INTERVENTIONS:
Other: inspiratory muscle training — Participants will complete inspiratory muscle training daily in their homes for 12 weeks. The dosage will depend on their initial maximum pressure. At the end of the 12 week intensive period, participants will reduce the inspiratory resistance by a third and continue a maintenance training for an additional 12 weeks.

SUMMARY:
People with PD have lower cardiopulmonary function than their age matched peers. This decline can further impair a person's ability to participate in exercise and daily activities.

Furthermore, the limitations in cardiopulmonary function can have a severe impact on mortality. There is evidence indicating the positive changes IMT can have on cardiopulmonary function in people with PD. Through intensive daily exercise people with PD have shown improvements in maximum inspiratory pressure and maximum expiratory pressure though detraining does occur when the intervention is not continued. The purpose of the proposed study is to determine if improvements in expiratory muscle strength can be maintained with a maintenance inspiratory muscle training program. The hypothesis is that there will be a significant change from baseline at the three and six month follow ups.

DETAILED DESCRIPTION:
Testers will complete the following outcome measures at the pretest: height, weight, maximum inspiratory pressure, maximum expiratory pressure, heart rate, blood pressure, respiratory rate, six-minute walk test, and Fatigue Impact Scale in person.17,18 Participants, and caregivers if necessary, will be educated on how to complete the intensive IMT program. The dosage will be IMT 3 times/day for 20 repetitions each with resistance set at 30% of baseline maximum for 12 weeks. This training will occur at home.

Participants will record daily their completion of the intensive IMT. Investigators will contact participants weekly for follow-up of compliance and questions. Participants will be contacted either through email, text, or phone call, depending on their preference.

After 12 weeks of intensive IMT training, the investigators will complete the first posttest which will include the following assessments: maximum inspiratory pressure, maximum expiratory pressure, heart rate, blood pressure, respiratory rate, six-minute walk test, and fatiguability scale in person.

Participants, and caregivers if necessary, will be educated on the maintenance IMT program. The dosage for the maintenance program will be 33% of their intensive IMT program, which will result in IMT 1 time/day for 20 repetitions with resistance set at 30% of baseline maximum at the first posttest. The participants will continue the maintenance program for 12 more weeks.

Participants will record daily their completion of the maintenance IMT program. Investigators will contact participants weekly for follow-up of compliance and questions. Participants will be contacted either through email, text, or phone call, depending on their preference.

After the 12 weeks of maintenance IMT, the investigators will complete the second posttest which will include the following assessments: maximum inspiratory pressure, maximum expiratory pressure, heart rate, blood pressure, respiratory rate, six-minute walk test, and fatiguability scale in person.

The participants will receive a $50 Amazon gift card upon the completion of second posttest. The participants will also be allowed to keep their IMT devices for continued use.

ELIGIBILITY:
Inclusion Criteria:

* physician's diagnosis of Parkinson's disease

Exclusion Criteria:

* people who are actively smoking, have a pacemaker, recent diagnosis of chronic obstructive pulmonary disease, bronchial asthma, active pulmonary disease within 1 month, or hospitalization within 2 months of time of study

Ages: 30 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
maximum expiratory pressure | 5 minutes
  measure of the maximum expiratory cardiopulmonary pressure
maximum inspiratory pressure | 5 minutes
  measure of the maximum inspiratory cardiopulmonary pressure
6 minute walk test | 8 minutes
  distance walked in 6 minutes
Fatigue Impact Scale | 10 minutes
  measure of a person's self report fatigue, ranges from 0-36 and higher score indicates greater impact of fatigue
heart rate | 1 minute
  heart beats per minutes
respiratory rate | 1 minute
  breaths per minute
blood pressure | 1 minute
  measure of rest blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Barta, PT, PhD, Principal Investigator — The University of St. Augustine for Health Sciences
Locations (1):
- University of St. Augustine for Health Sciences, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No